CLINICAL TRIAL: NCT05809167
Title: Venetoclax (VEN)+Azacytidine (AZA) Followed by Modified BUCY Conditioning Regimen for High Risk or Refractory/Relapsed Acute Lymphoblastic Leukemia Undergoing Allogeneic Hematopoietic Stem Cell Transplantation (Allo-HSCT)
Brief Title: Venetoclax+Azacytidine+Modified BUCY Conditioning Regimen for Acute Lymphoblastic Leukemia Undergoing Allo-HSCT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VA+mBUCY-02
Record Dates: First submitted 2023-02-27; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-02

CONDITIONS: Allogeneic Hematopoietic Stem Cell Transplantation; Acute Lymphoblastic Leukemia
Keywords: venetoclax; azacytidine; hematopoietic stem cell transplantation; acute lymphoblastic leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VEN+AZA+Modified BUCY (Experimental)
  Interventions: Drug: VEN+AZA+Modified BUCY

INTERVENTIONS:
Drug: VEN+AZA+Modified BUCY — Venetoclax: 200mg/day*7days（It should be combined with triazole antifungal drugs).
  Azacytidine: 75mg/ m²/day*7days.

SUMMARY:
The purpose of this prospective, open-label, single-center study is to evaluate the efficacy and safety of VEN-AZA (venetoclax and azacytidine) followed by modified BUCY (busulfan and cyclophosphamide) as conditioning regimen for high-risk or relapsed/refractory acute lymphoblastic leukemia (ALL) undergoing allogeneic hematopoietic stem cell transplantation (allo-HSCT).

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (Allo-HSCT) is the only potentially curative therapy for patients with acute lymphoblastic leukemia. However, relapse remains a leading cause for treatment failure after hematopoietic cell transplantation (HCT) in patients, optimization of conditioning regimen can improve prognosis and decrease relapse. Abnormal gene methylation is common in ALL patients. Azacytidine is a DNA methylation transferase inhibitor that can re-express tumor suppressor genes in leukemia cells. Venetoclax is a selective BCL-2 inhibitor, which has antitumor activity against a variety of hematological malignancies. The combination of the two drugs show a synergistic anti-tumor effect. Multiple case reports the efficacy of Venetoclax-based regimens in patients with ALL is encouraging. The objective of this study is to evaluate the feasibility, safety and efficacy of VEN-AZA bridging allogeneic hematopoietic stem cell transplantation in the treatment of high-risk ALL.

ELIGIBILITY:
Inclusion Criteria:

1. Age 14 to 65 years;
2. Diagnosis of high-risk or relapsed/refractory acute lymphoblastic leukemia at the time of transplant.
3. Must need a bone marrow transplant;
4. Must have the ability to observe the efficacy and events;
5. Patient must have ability to understand and willingness to provide written informed consent prior to participation in the study and any related procedures being performed.

Exclusion Criteria:

1. Age <14 or >65 years;
2. Uncontrolled bacterial, viral, fungal, or other infection before conditioning regimen;
3. Pregnant or lactating females;
4. Current participation in another clinical trial;
5. Contra-indication to one of the drug of the regimen;
6. Any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney, liver or other organ system that may place the patient at undue risk to undergo the agents included in the conditioning regimen

Ages: 8 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2025-01-20 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
disease-free survival (DFS) | 3 years after transplantation
  It is measured from the time from randomization to the first of relapse or death.
overall survival (OS) | 3 years after transplantation
  It is measured from the time of entry into this trial to the date of death from any cause; patients not known to have died at last follow-up are censored on the date they were last known to be alive.

SECONDARY OUTCOMES:
veno-occlusive disease (VOD) | 3 years after transplantation
  incidence of veno-occlusive disease (VOD) events (refer to modified Seattle Criteria of VOD)
graft-versus-host disease (GvHD) | 3 years after transplantation
  incidence and severity of acute (aGvHD) and chronic graft-versus-host disease (cGvHD) (aGvHD refer to Glucksberg Criteria and cGvHD refer to the National Institutes of Health Consensus)
transplant related mortality (TRM) | 3 years after transplantation
  cumulative incidence of transplant related mortality
Regimen related toxicity | 3 years after transplantation
  Number of participants with regimen related toxicity as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Depei Wu Wu, MD, Study Chair — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No